CLINICAL TRIAL: NCT00875693
Title: A Novel Sequential Treatment of Salvage and Reduced Intensity Conditioning RIC) Chemotherapy for Allogeneic Stem-Cell Transplantation (SCT)for Primary Refractory and Relapsed Acute Myelogenous Leukemia
Brief Title: A Novel Sequential Treatment of Salvage and Reduced Intensity Conditioning (RIC) Chemotherapy for Allogeneic Stem-Cell Transplantation (SCT) for Primary Refractory and Relapsed Acute Myelogenous Leukemia (AML)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0812010140
Record Dates: First submitted 2009-04-02; First posted 2009-04-03 (Estimated); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Acute Myelogenous Leukemia; Myelodysplastic Syndrome
Keywords: AML; leukemia; MDS
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Leukemia | interventions — CPX-351

ARMS (2):
- Arm A dose of CPX - 351 (Experimental): Dose level 1A: 60 units/m2 days -28, -26 and -24 Dose level 2A: 80 units/m2 days -28, -26 and -24 Dose level 3A: 100 units/m2 days -28, -26 and -24 Dose level 4A: 120 units/m2 days -28, -26 and -24 Dose level 5A: 140 units/m2 days -28, -26 and -24 Dose level 6A: 160 units/m2 days -28, -26 and -24
  Interventions: Drug: CPX-351
- Arm B dose of CPX-351 (Experimental): Dose level 1B: 60 units/m2 days -21, -19 and -17 Dose level 2B: 80 units/m2 days -21, -19 and -17 Dose level 3B: 100 units/m2 days -21, -19 and -17 Dose level 4B: 120 units/m2 days -21, -19 and -17 Dose level 5B: 140 units/m2 days -21, -19 and -17
  Interventions: Drug: CPX-351

INTERVENTIONS:
Drug: CPX-351 — CPX-351 is a liposomal formulation of a fixed combination of the antineoplastic drugs cytarabine and daunorubicin. The two drugs are present inside the liposome in a 5:1 molar ratio.

SUMMARY:
This open-label Phase I study is designed to determine the maximum tolerated dose (MTD) for CPX-351 followed by a reduced intensity conditioning regimen and incorporates a dose-escalation schedule that sequentially enrolls 6 dosing cohorts. After the determination of the MTD, the investigator reserves the option to enroll up to 10 additional subjects in an expanded safety cohort(s) at the MTD.

Refractory and relapsed AML patients who meet standard institutional criteria to undergo sequential induction/reduced intensity conditioning allogeneic transplants will be offered a transplant from a related or unrelated donor (full match or 1 antigen mismatch). Cord blood transplants will not be used in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients are included, if they fulfill at least one of the following criteria defining refractory or relapsed AML according to previously established criteria 1-3: (1) Primary induction failure (PIF) after ≥ 2 cycles of chemotherapy. (2) First relapse. (3) Relapse refractory to salvage chemotherapy (4) Second or subsequent relapse.
2. Patients with MDS, either refractory anemia with excess blasts (RAEB) I or RAEB II
3. Age between 18 and 70 years old.
4. Patients must have a Karnofsky Performance Status > 70.
5. Each patient must be willing to participate as a research subject and must sign an informed consent form.
6. If the patient has a history of a prior malignancy, they must be without any evidence of disease of that prior malignancy for at least 2 years before being eligible for transplant on this protocol. This excludes skin cancers that may have been excised within that 2 year period.
7. Patients must have adequate physical function measured by:

   1. Cardiac: asymptomatic or if symptomatic then left ventricular ejection fraction (LVEF) at rest must be > 50% and must improve with exercise.
   2. Hepatic: < 3x upper limit of normal (ULN) alanine aminotransferase (ALT) and < 1.5 total serum bilirubin, unless liver is involved with the disease or there is congenital benign hyperbilirubinemia.
   3. Renal: serum creatinine within normal range for age or if serum creatinine is outside the normal range, then creatinine clearance > 60-ml/min.
   4. Pulmonary: asymptomatic or if symptomatic, diffusing capacity of carbon monoxide (DLCO) > 45% of predicted (corrected for hemoglobin)

Exclusion Criteria:

1. Impaired renal function with a measured or calculated creatinine clearance of less than 60 ml/min.
2. Impaired hepatic function defined as a bilirubin greater than 1.5 x upper limit of normal or alanine aminotransferase (ALT) or aspartate aminotransferase (AST) greater than 3 x normal.
3. Serious active or uncontrolled infection (Infections are controlled when patients are afebrile and hemodynamically stable for 72 hours) or medical condition.
4. Women who are pregnant or breast feeding. Women of childbearing age must use adequate contraception and have a negative pregnancy test.
5. Impaired pulmonary function with a DLCO less than 45% predicted.
6. Impaired cardiac function with an ejection fraction less than 50% of predicted by echocardiogram or multigated acquisition scan (MUGA).
7. Prior daunorubicin therapy with a cumulative dose of more than 368 mg/m2 or equivalent. The anthracycline agents commonly used in treating myeloid malignancies are doxorubicin, idarubicin and mitoxantron.

   For example, a patient who receives 7 + 3 (daunorubicin 180 mg/m2) for induction and MEC regimen (mitoxantrone, etoposide, cytaragine; mitoxantrone 48 mg/m2) for salvage. The cumulative daunorubicin equivalent is 180 + (48x2) = 278 mg/m2.
8. Other systemic anticancer therapy or ongoing toxicities from such therapy.
9. Patients with a history of and/or current evidence of myocardial impairment (e.g. cardiomyopathy, ischemic heart disease, significant valvular dysfunction, hypertensive heart disease, congestive heart failure), resulting in heart failure by New York Heart Association Class III or IV staging.
10. Patients with Wilson disease or other Copper-related disorders.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2009-06-02 (Actual); Primary Completion 2014-06-30 (Actual); Study Completion 2017-12-27 (Actual)

PRIMARY OUTCOMES:
To determine the toxicity and safety of the regimen | cohort dependent

CONTACTS AND LOCATIONS:
Overall Officials: Usama Gergis, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States